CLINICAL TRIAL: NCT05876221
Title: Platelet Response to Caplacizumab in the Treatment of Acquired Thrombotic Thrombocytopenic Purpura
Acronym: PREDICT2020
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Paul Brinkkoetter, Consultant in Nephrology, University of Cologne
Other Study IDs: 2020-11-17
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
Keywords: caplacizumab; platelet responses; aTTP; iTTP
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aTTP-Patients: Patients with immune Thrombotic Thrombocytopenic Purpura, who have been treated with caplacizumab (Cablivi®)
  Interventions: Drug: Cablivi

INTERVENTIONS:
Drug: Cablivi — Patients with immune Thrombotic Thrombocytopenic Purpura, who have been treated with caplacizumab (Cablivi®)

SUMMARY:
The interpretation of platelet counts has to be revaluated in the light of caplacizumab. By effectively blocking platelet binding sites on VWF-multimers, the nanobody leads to a rapid normalization of the platelet count within 3 to 4 days. Most importantly, caplacizumab uncouples platelet counts from ADAMTS13 activity and thereby launches unprecedented thrombocyte dynamics, with potential pitfalls for over- and undertreatment.

A relevant number of patients responds to caplacizumab with a brisk increase in platelet count, followed by a marked dip of platelets (patient on the left). This may mislead treating physicians into re-intensifying therapy, with a respective risk for adverse side-effects and complications. Taken together, these observations call for reliable descriptions and the identification of predictive parameters to predict the platelet response upon administration of caplacizumab in a large patient cohort. Here, PREDICT-2020 is designed as a retrospective study to specifically address the following aspects:

* Identifying and describing clusters of platelet responses to caplacizumab
* Identifying potential pitfalls for treating physicians
* Predicting the individual thrombocyte response
* Correlating platelet responses with individual patient outcome

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autoimmune thrombotic thrombocytopenic purpura
* Treatment with at least a single dose of caplacizumab, either i.v. or s.c.
* Male or female patients older than 18 years of age

Exclusion Criteria:

* Hereditary thrombotic thrombocytopenic purpura

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this trial will be enclosed iTTP patients treated with caplacizumab from:
  * the German real-world cohort of iTTP patients treated with caplacizumab in the years 2018 to 2020 , and
  * the respective TITAN and HERCULES trial cohorts.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Reliable description and prediction of platelet responses to caplacizumab | Enrollment
  Reliable description and prediction of platelet responses to caplacizumab employing mathematic modelling algorithms

SECONDARY OUTCOMES:
Determination of different clusters of platelet responses to caplacizumab | Enrollment
  It will be hypothesized the existence of different clusters of caplacizumab responders during the first weeks of therapy, when ADAMTS13 activity typically is still <10%. A detailed cluster analysis and description of thrombocyte responses to caplacizumab in a large cohort will reliably identify these different responders
Correlation of platelet responses to caplacizumab with patient outcome | Enrollment
  It will be hypothesized the existence of different clusters of caplacizumab responders during the first weeks of therapy, when ADAMTS13 activity typically is still <10%. A detailed cluster analysis and description of thrombocyte responses to caplacizumab in a large cohort will reliably identify these different responders
Risk stratification of iTTP patients based on their platelet response to caplacizumab | Enrollment
  Description: Predicting the individual thrombocyte response to caplacizumab improves risk stratification of iTTP patients after initiation of caplacizumab therapy. An early risk stratification allows an optimal timing of monitoring intervals during the first weeks after diagnosis, which are often critical

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Kühne, MD, Principal Investigator — Department II of Internal Medicine, University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany